CLINICAL TRIAL: NCT03157726
Title: Transurethral Plasmakinetic Enucleation of Prostate Versus Transurethral Resection of Prostate: A Multi-center Randomized Control Trial
Brief Title: Transurethral Plasmakinetic Enucleation of Prostate Versus Transurethral Resection of Prostate
Acronym: ERP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Fourth Affiliated Hospital of Guangxi Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC2016ZD025
Record Dates: First submitted 2017-05-11; First posted 2017-05-17 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; multicenter randomized control clinical trial; transurethral plasmakinetic enucleation of prostate; transurethral resection of prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUKEP(enucleation of prostate) (Active Comparator): Patients accept TUKEP (transurethral plasmakinetic enucleation of prostate). The TUKEP procedure requires the use of a resectoscope, camera system and irrigation fluid. The system consists of a generator unit and a wire loop with an electrical current running, the beak of resectoscope was used to enucleation of prostate and the bipolar loop was used to cutting and coagulation, There are many manufacturers of Bipolar TURP systems. Any bipolar plasmakinetic system approved by the CFDA (Chinese food and drug administration) may be used for the study.
  The bipolar plasmakinetic system was set at 160 W for cutting and 100 W for coagulation.
  Interventions: Procedure: Transurethral plasmakinetic enucleation of prostate
- TURP(resection of prostate) (Active Comparator): Patients accept TURP (transurethral resection of prostate). The TURP procedure requires the use of a resectoscope, camera system and irrigation fluid. The system consists of a generator unit and a wire loop with an electrical current running through the loop used to cut prostate tissue and cauterize. Prostate tissue is cut away in small pieces and removed at the end of the procedure using irrigation. There are many manufacturers of TURP systems. Any monopolar and bipolar loop system approved by the CFDA (Chinese food and drug administration) may be used for the study.
  The bipolar plasmakinetic system was set at 160 W for cutting and 100 W for coagulation.
  Interventions: Procedure: transurethral resection of prostate

INTERVENTIONS:
Procedure: Transurethral plasmakinetic enucleation of prostate — Transurethral plasmakinetic enucleation of prostate(PAKEP),an operation mode devised by Liu Chunxiao Team in southern medical university urology department. The theory of the operation is using transurethral resectoscope instead of the finger in the open operation, to find the surgical capsule of prostate and to peel the hyperplastic prostate gland visually in a antidromic way.
  Other Names: TUKEP
  Arms: TUKEP(enucleation of prostate)
Procedure: transurethral resection of prostate — Transurethral resection of prostate(TURP), a kind of mature minimally invasive surgery of prostate , taking the place of the traditional open surgery in 1930s , still is the "gold standard" operation for surgical treatment of BPH.
  Other Names: TURP
  Arms: TURP(resection of prostate)

SUMMARY:
The study is a multicentric randomized control trial with 4-year follow-up comparing perioperative and postoperative outcomes for transurethral plasmakinetic enucleation of prostate(TUKEP) and transurethral resection of prostate(TURP). The investigators recruit patient with benign prostatic hyperplasia(BPH) as the object of study. TURP is set as control group . Meanwhile TUKEP is set as test group. Six affiliated hospitals will participate in this study. Through analyzing the perioperative and postoperative data between TUKEP group and TURP group, The investigators purpose demonstrating superiority of safety, efficacy and economic benefit in TUKEP group.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is the most common disease of middle aged and elderly people which cause urinary tract symptoms (LUTS). transurethral resection of prostate(TURP) , began to replace the traditional open surgery in 1930s, still is as the "gold standard" operation for surgical treatment of BPH. However, compared with the traditional open operation, TURP has the following flaws:(1), due to the incomplete resection , maximum flow rate(Qmax) after TURP is lower than Qmax after open surgery. (2), there are serious complications, such as water intoxication and hemorrhage. (3) TURP has limitation to large prostate.

Transurethral plasmakinetic enucleation of prostate(TUKEP), an operation mode devised by Liu Chunxiao Team in southern medical university urology department, have offset the advantage of TURP. The theory of the operation is using transurethral resectoscope instead of the finger in the open operation, to find the surgical capsule of prostate and to peel the hyperplastic prostate gland visually in a antidromic way. One the one hand, TUKEP effectively solve the situation that It should repeatedly cut and stop bleeding and difficultly find the surgical capsule in TURP, which obviously reduce the rate of bleeding, prostatic capsula perforation, transurethral resection syndrome(TURS) and External sphincter injury. On the other hand, TUKEP is the minimally invasive surgery. It also achieves the effect of open surgery resolving the residual gland and reoperation post TURP.

The investigators plan to setup a a multicentric randomized control trial with 4-year follow-up comparing perioperative and postoperative outcomes for TUKEP and TURP. Through analyzing the perioperative and postoperative data between TUKEP group and TURP group, The purpose demonstrating superiority of safety, efficacy and economic benefit in TUKEP group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose as BPH
2. Between 50 and 80 year-old
3. Prostate volume less than 120g
4. Meet any conditions (1). International Prostate Symptom Score (IPSS),≥12 quality of life score (QOL) ≥4分 (2).Maximum urinary flow rate (Qmax) 15 ml/s or less (urine flow more than 150 ml) (3).Medication is not efficient (4).Repeated urinary retention (extubation failure more than one) (5).Schafer≥grade 2
5. The American association of anesthesia score (ASA) class 1 to 3
6. Sign the informed consent voluntarily and will be willing to follow-up

Exclusion Criteria:

1. Combined with central nervous system lesions (such as cerebrovascular accident, Parkinson, multiple sclerosis, cauda equina injury, spinal cord lesions, etc.) and neurogenic bladder;
2. The combination of advanced malignant tumor or chronic wasting disease;
3. Patients with severe cardiopulmonary disease or severe mental disorders;
4. Acute urinary tract infection, urethral stricture;
5. There is a history of prostate and bladder surgery;
6. Combined with severe coagulopathy;
7. Postoperative pathology confirmed prostate cancer;
8. Poor compliance, and can not be followed up.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-06-06 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Qmax(Maximum urinary flow rate) | 4 years
  Maximum urinary flow rate was measured at 1, 3, 6, 12, 24, 36 and 48-month postoperatively
IPSS (International Prostate Symptom Score ) | 4 years
  International Prostate Symptom Score was measured at 1, 3, 6, 12, 24, 36 and 48-month postoperatively

SECONDARY OUTCOMES:
QOL(Quality of Life) | 4 years
  The Quality of Life Score was measured at 1, 3, 6, 12, 24, 36 and 48-month postoperatively
International Index Of Erectile Function (IIEF-5) | 4 years
  International Index Of Erectile Function is a patient reporting outcomes measuring the erectile function at the baseline, 1,3,6,12, 24,36 and 48-month follow-up visits postoperatively.
Operation time | up to 24 hours
  operation time
Postoperative hospital stay | 1 month
  Postoperative hospital stay
Indwelling catheter time | 1 month
  The time of indwelling catheter post-operation
Postoperative irrigation | 1 month
  The time of Postoperative irrigation
Decrease in Haemoglobin in 24 hours post-operation | 1 month
  Compared with the baseline, to demonstrate the blood loss during operation
Retreatment rate | 4 years
  The ratio of patient who need reoperation to remove urinary tract obstruction
Prostate-specific antigen(PSA) | 4 years
  To compare the Prostate-specific antigen between TUKEP and TURP at baseline, 1,3,6,12, 24,36 and 48-month follow-up visits.
Hospitalization expenses | 1 month
  Total costs for BPH treatment during Hospitalization. The cost of other diseases should be excluded
Prostate volume | 4 years
  Prostate volume is measured by ultrasound or MRI at the baseline, 1,3,6,12, 24,36 and 48-month follow-up visits
Residual urine volume | 4 years
  Residual urine in the bladder after urination(via abdominal ultrasonography) is measure at the baseline, 1,3,6,12, 24,36 and 48-month follow-up visits
Claviendindo classification | 4 years
  It is a grade for evaluating surgical complications at 1,3,6,12, 24,36 and 48-month follow-up visits

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No